CLINICAL TRIAL: NCT03833427
Title: A Phase 1b Multi-center Clinical Study of Selumetinib (MK-5618) in Combination With Pembrolizumab (MK-3475) in Participants With Advanced/Metastatic Solid Tumors.
Brief Title: Study of Selumetinib (MK-5618) in Combination With Pembrolizumab (MK-3475) in Participants With Advanced/Metastatic Solid Tumors (MK-5618-001)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 5618-001; MK-5618-001 (Other: MSD Protocol Number)
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Advanced/Metastatic Solid Tumors
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — AZD 6244; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Selumetinib at Dose Level 1 + Pembrolizumab (Experimental): Participants receive 200 mg pembrolizumab (IV infusion; every three weeks [Q3W]) in combination with selumetinib at dose level 1 (dosed orally; twice daily [BID]) for up to 35 treatment cycles (cycle length: 3 weeks). During each 3-week cycle, selumetinib will be administered only for the first two weeks.
  Interventions: Drug: Selumetinib; Drug: Pembrolizumab
- Selumetinib at Dose Level 2 + Pembrolizumab (Experimental): Participants receive 200 mg pembrolizumab (IV infusion; Q3W) in combination with selumetinib at dose level 2 (dosed orally; BID) for up to 35 treatment cycles (cycle length: 3 weeks). During each 3-week cycle, selumetinib will be administered only for the first two weeks.
  Interventions: Drug: Selumetinib; Drug: Pembrolizumab
- Selumetinib at Dose Level 3 + Pembrolizumab (Experimental): Participants receive 200 mg pembrolizumab (IV infusion; Q3W) in combination with selumetinib at dose level 3 (dosed orally; BID) for up to 35 treatment cycles (cycle length: 3 weeks). During each 3-week cycle, selumetinib will be administered only for the first two weeks.
  Interventions: Drug: Selumetinib; Drug: Pembrolizumab
- Selumetinib at Dose Level 4 + Pembrolizumab (Experimental): Participants receive 200 mg pembrolizumab (IV infusion; Q3W) in combination with selumetinib at dose level 4 (dosed orally; BID) for up to 35 treatment cycles (cycle length: 3 weeks). During each 3-week cycle, selumetinib will be administered only for the first two weeks.
  Interventions: Drug: Selumetinib; Drug: Pembrolizumab
- Selumetinib at Dose Level 5 + Pembrolizumab (Experimental): Participants receive 200 mg pembrolizumab (IV infusion; Q3W) in combination with selumetinib at dose level 5 (dosed orally; BID) for up to 35 treatment cycles (cycle length: 3 weeks). During each 3-week cycle, selumetinib will be administered only for the first two weeks.
  Interventions: Drug: Selumetinib; Drug: Pembrolizumab
- Selumetinib at Dose Level 6 + Pembrolizumab (Experimental): Participants receive 200 mg pembrolizumab (IV infusion; Q3W) in combination with selumetinib at dose level 6 (dosed orally; BID) for up to 35 treatment cycles (cycle length: 3 weeks). During each 3-week cycle, selumetinib will be administered only for the first two weeks.
  Interventions: Drug: Selumetinib; Drug: Pembrolizumab
- Selumetinib at Dose Level 7 + Pembrolizumab (Experimental): Participants receive 200 mg pembrolizumab (IV infusion; Q3W) in combination with selumetinib at dose level 7 (dosed orally; BID) for up to 35 treatment cycles (cycle length: 3 weeks). During each 3-week cycle, selumetinib will be administered only for the first two weeks.
  Interventions: Drug: Selumetinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Selumetinib — Selumetinib oral capsules administered BID at escalating dose levels. Selumetinib administered only in weeks 1&2 of each 3-week treatment cycle.
  Other Names: MK-5618
Drug: Pembrolizumab — Pembrolizumab administered by IV infusion at 200 mg Q3W, given on cycle day 1 of each 3-week treatment cycle.
  Other Names: KEYTRUDA®; MK-3475

SUMMARY:
This study will examine the safety, pharmacokinetics, and efficacy of escalating doses of selumetinib (MK-5618) in combination with intravenous (IV) pembrolizumab (MK-3475) for participants with advanced / metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed advanced or metastatic solid tumor by pathology report and have received, or been intolerant to, all treatment known to confer clinical benefit.
* Has measurable disease by Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1) as assessed by local site investigator/radiology. Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Is able to swallow and retain oral medication and has no clinically significant gastrointestinal abnormalities that might alter absorption.
* Has adequate organ function.
* If male, agree to use a contraception during the treatment period and for at least 120 days after the last dose of study intervention and refrain from donating sperm during this period.
* If female, is not pregnant or breastfeeding, and is not a woman of childbearing potential (WOCBP). If a WOCBP, agree to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study intervention.
* For Human immunodeficiency virus (HIV) infected participants, must have well controlled HIV on a stable regimen of anti-retroviral therapy (ART). Participants on ART must have been without changes in drugs or dose modification for at least 4 weeks prior to study entry.

Exclusion Criteria:

* Has had chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks (2 weeks for palliative radiation) prior to the first dose of study treatment, or has not recovered to Common Toxicity Criteria for Adverse Events (CTCAE) Grade 1 or better from any AEs that were due to cancer therapeutics administered more than 4 weeks earlier (this includes participants with previous immunomodulatory therapy with residual immune-related AEs). Participants receiving ongoing replacement hormone therapy for endocrine immune-related AEs will not be excluded from participation in this study.
* Has clinically active central nervous system metastases and/or carcinomatous meningitis.
* Has had a severe hypersensitivity reaction (≥ Grade 3) to treatment with a monoclonal antibody/component of the study treatment, and/or has a history of allergic reactions attributed to compounds of similar chemical or biologic composition to agents and/or excipients used in the study.
* Has an active infection requiring therapy.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years except vitiligo or resolved childhood asthma/atopy. Replacement therapy, such as thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, is not considered a form of systemic treatment and is allowed. Use of non-systemic steroids is permitted.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to allocation.
* Has known Hepatitis B or C infection.
* For HIV infected participants, has a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
* Has undergone major surgery and has not recovered adequately from any toxicity and/or complications from the intervention prior to starting study therapy.
* Has baseline peripheral neuropathy/paresthesia Grade 1.
* Has any medical, psychiatric, cognitive, or other condition that may compromise the participant's ability to understand the participant information, give informed consent, comply with the study protocol, or complete the study, in the opinion of the treating investigator.
* Participants with clinically significant cardiovascular disease as defined by the following: 1) Uncontrolled hypertension; 2) Left ventricular ejection fraction (LVEF) <55%; 3) Symptomatic heart failure (New York Heart Association (NYHA) Grade II to IV), prior or current cardiomyopathy, or severe valvular heart disease; 4) Uncontrolled angina; 5) Clinically significant cardiac arrhythmia and/or conduction abnormality ≤6 months prior to start of study treatment; 6) Myocardial infarction or acute coronary syndrome ≤6 months prior to start of study treatment; 7) Mean QT interval calculated according to the Frederica method (QTcF) interval: Male >450 ms; Female >470 ms.
* Has a history of thromboembolic or cerebrovascular event(s) within 6 months prior to study enrollment, including transient ischemic attack, cerebrovascular accident, deep vein thrombosis, or pulmonary embolism.
* Has a neuromuscular disorder associated with an elevated creatine kinase (e.g., inflammatory myopathy, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy.
* Has a history of, or current, retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma, ocular hypertension, history of hyperviscosity, or hypercoagulability syndromes).
* Has retinal degenerative disease.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, make administration of the study treatments hazardous or make it difficult to monitor adverse effects such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has a known psychiatric or substance abuse disorder that would interfere with the Participant's ability to cooperate with the requirements of the study.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
* Has received a live-virus vaccine within 28 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.
* Is currently participating and receiving study treatment in a study of an investigational agent or has participated and received study treatment in a study of an investigational agent or has used an investigational device within 28 days of administration of selumetinib.
* Is a WOCBP who has a positive urine pregnancy test within 24 hours before the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (6):
- United States (4):
  - City of Hope National Medical Center ( Site 0004), Duarte, California
  - START Midwest ( Site 0001), Grand Rapids, Michigan
  - John Theurer Cancer Center ( Site 0002), Hackensack, New Jersey
  - South Texas Accelerated Research Therapeutics, LLC (START) ( Site 0003), San Antonio, Texas
- Canada (2):
  - Princess Margaret Cancer Centre ( Site 0014), Toronto, Ontario
  - CHU de Quebec Universite de Laval ( Site 0013), Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Chenard-Poirier M, Hansen AR, Gutierrez ME, Rasco D, Xing Y, Chen LC, Zhou H, Webber AL, Freshwater T, Sharma MR. A phase 1 trial of the MEK inhibitor selumetinib in combination with pembrolizumab for advanced or metastatic solid tumors. Invest New Drugs. 2024 Jun;42(3):241-251. doi: 10.1007/s10637-024-01428-0. Epub 2024 Mar 14. PMID 38483782
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Though the total planned enrollment for this study was 50 participants. Only 32 participants were allocated and included in Part 1, dose escalation for analysis. Part 2 cohort expansion was not initiated. The study was terminated after completion of dose escalation due to reasons unrelated to safety or tolerability.
Groups:
- Selumetinib 50mg + Pembrolizumab: Participants received 200 mg pembrolizumab (IV infusion; every three weeks [Q3W]) in combination with selumetinib 50mg orally twice daily [BID]) for up to 35 treatment cycles (cycle length: 3 weeks). During each 3-week cycle, selumetinib was administered only for the first two weeks.
- Selumetinib 75mg + Pembrolizumab: Participants received 200 mg pembrolizumab (IV infusion; every three weeks [Q3W]) in combination with selumetinib 75mg orally twice daily [BID]) for up to 35 treatment cycles (cycle length: 3 weeks). During each 3-week cycle, selumetinib was administered only for the first two weeks.
- Selumetinib 100mg + Pembrolizumab: Participants received 200 mg pembrolizumab (IV infusion; every three weeks [Q3W]) in combination with selumetinib 100mg orally twice daily [BID]) for up to 35 treatment cycles (cycle length: 3 weeks). During each 3-week cycle, selumetinib was administered only for the first two weeks.
- Selumetinib 125mg + Pembrolizumab: Participants received 200 mg pembrolizumab (IV infusion; every three weeks [Q3W]) in combination with selumetinib 125mg orally twice daily [BID]) for up to 35 treatment cycles (cycle length: 3 weeks). During each 3-week cycle, selumetinib was administered only for the first two weeks.
- Selumetinib 150mg + Pembrolizumab: Participants received 200 mg pembrolizumab (IV infusion; every three weeks [Q3W]) in combination with selumetinib 150mg orally twice daily [BID]) for up to 35 treatment cycles (cycle length: 3 weeks). During each 3-week cycle, selumetinib was administered only for the first two weeks.
- Selumetinib 200mg + Pembrolizumab: Participants received 200 mg pembrolizumab (IV infusion; every three weeks [Q3W]) in combination with selumetinib 200mg orally twice daily [BID]) for up to 35 treatment cycles (cycle length: 3 weeks). During each 3-week cycle, selumetinib was administered only for the first two weeks.
- Selumetinib Above 200mg (up to 300mg) + Pembrolizumab: Participants received 200 mg pembrolizumab (IV infusion; every three weeks [Q3W]) in combination with selumetinib above 200mg (up to 300mg) orally twice daily [BID]) for up to 35 treatment cycles (cycle length: 3 weeks). During each 3-week cycle, selumetinib was administered only for the first two weeks.
Period: Overall Study
Arm/Group | Selumetinib 50mg + Pembrolizumab | Selumetinib 75mg + Pembrolizumab | Selumetinib 100mg + Pembrolizumab | Selumetinib 125mg + Pembrolizumab | Selumetinib 150mg + Pembrolizumab | Selumetinib 200mg + Pembrolizumab | Selumetinib Above 200mg (up to 300mg) + Pembrolizumab
Started | 4 | 3 | 11 | 14 | 0 | 0 | 0
Discontinued | 4 | 3 | 11 | 14 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 11 | 14 | 0 | 0 | 0
Not completed — Death | 4 | 2 | 9 | 11 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 1 | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Selumetinib 50mg + Pembrolizumab | Selumetinib 75mg + Pembrolizumab | Selumetinib 100mg + Pembrolizumab | Selumetinib 125mg + Pembrolizumab | Total
Number analyzed (Participants) | 4 | 3 | 11 | 14 | 32
Age, Customized [Number; unit: Participants]
  Between 18 and 64 years | 4 | 3 | 10 | 12 | 29
  From 65 to 84 years | 0 | 0 | 1 | 2 | 3
  85 years and over | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 3 | 10
  Male | 2 | 2 | 7 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 4 | 5
  Not Hispanic or Latino | 4 | 1 | 11 | 10 | 26
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 9 | 11 | 27
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose-Limiting Toxicities (DLTs)
Description: DLT was defined as toxicities that: 1) were possibly, probably, or definitely related to study therapy, excluding toxicities clearly not related to the drug, such as disease progression, environmental factors, unrelated trauma; and 2) met pre-defined severity criteria. For each arm, the number of participants experiencing DLTs were assessed.
Time Frame: Up to 21 days
Population: All allocated participants who received at least one dose of study treatment and met the protocol-specified criteria for DLT evaluability.
Measure: Count of Participants; unit: Participants
Arm/Group | Selumetinib 50mg + Pembrolizumab | Selumetinib 75mg + Pembrolizumab | Selumetinib 100mg + Pembrolizumab | Selumetinib 125mg + Pembrolizumab
Number analyzed (Participants) | 2 | 3 | 11 | 14
Participants | 0 | 0 | 2 | 3

2. Primary Outcome: Number of Participants Who Experienced Adverse Event (AE)
Description: An AE was any unfavorable and unintended sign, symptom, or disease (new or exacerbated) in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. For each arm, the number of participants experiencing an AE will be assessed.
Time Frame: Up to ~28 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Selumetinib 50mg + Pembrolizumab | Selumetinib 75mg + Pembrolizumab | Selumetinib 100mg + Pembrolizumab | Selumetinib 125mg + Pembrolizumab
Number analyzed (Participants) | 4 | 3 | 11 | 14
Participants | 4 | 3 | 11 | 14

3. Primary Outcome: Number of Participants Discontinuing Study Treatment Due to an Adverse Event
Description: An AE was any unfavorable and unintended sign, symptom, or disease (new or exacerbated) in a clinical study participant, temporally associated withthe use of study treatment, whether or not considered related to the study treatment. For each arm, the number of participants discontinuing study treatment due to an AE was assessed.
Time Frame: Up to ~28 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Selumetinib 50mg + Pembrolizumab | Selumetinib 75mg + Pembrolizumab | Selumetinib 100mg + Pembrolizumab | Selumetinib 125mg + Pembrolizumab
Number analyzed (Participants) | 4 | 3 | 11 | 14
Participants | 0 | 1 | 4 | 3

4. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) of Selumetinib.
Description: Plasma selumetinib concentration was quantified for each arm to determine AUC, defined as the area under the concentration-time curve for selumetinib. AUC(0-last) is area under the concentration-time curve from dosing (time 0) to the time of the last measured concentration. AUC (0-12) is area under the concentration-time curve from dosing (time 0) to 12 hours.
Time Frame: Pre-dose, 1, 2, 4, 6, between 8 and 12 hours post dose on Day 1; Time 0 pre-dose at Cycle 2 Day 1, Cycle 2 Day 14, Cycle 5 Day 1 and Cycle 5 Day 14.
Population: All allocated participants who were compliant with the study procedures and had AUC data available from at least 1 treatment dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Selumetinib 50mg + Pembrolizumab | Selumetinib 75mg + Pembrolizumab | Selumetinib 100mg + Pembrolizumab | Selumetinib 125mg + Pembrolizumab
Number analyzed (Participants) | 4 | 3 | 11 | 14
hr*ng/mL
  AUC0-last | 2080 (71.4) | 3800 (5.7) | 4660 (51.2) | 4430 (57.6)
  AUC0-12 | 2160 (73.1) | 4220 (8.5) | 5060 (47.7) | 4760 (62.0)

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Selumetinib
Description: Plasma selumetinib concentration was quantified for each arm to determine Cmax, defined as the maximum observed concentration of selumetinib in plasma.
Time Frame: as for outcome 4
Population: All allocated participants who were compliant with the study procedures and had Cmax data available from at least 1 treatment dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Selumetinib 50mg + Pembrolizumab | Selumetinib 75mg + Pembrolizumab | Selumetinib 100mg + Pembrolizumab | Selumetinib 125mg + Pembrolizumab
Number analyzed (Participants) | 4 | 3 | 11 | 14
ng/mL | 852 (79.5) | 1400 (33.4) | 1690 (90.4) | 1410 (70.5)

6. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of Selumetinib
Description: Plasma selumetinib concentration was quantified for each arm to determine Cmin, defined as the minimum observed concentration of selumetinib in plasma.
Time Frame: as for outcome 4
Population: All allocated participants who were compliant with the study procedures and had Cmin data available from at least 1 treatment dose at each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: %GCV
Arm/Group | Selumetinib 50mg + Pembrolizumab | Selumetinib 75mg + Pembrolizumab | Selumetinib 100mg + Pembrolizumab | Selumetinib 125mg + Pembrolizumab
Number analyzed (Participants) | 2 | 3 | 7 | 12
%GCV
  Selumetinib-Cycle 2 Day 1 | NA (NA) — NA=Geometric Mean (%GCV) were not calculated due to all Selumetinib plasma concentrations were below the level of detection at Cycle 2 Day 1. | NA (NA) — NA=Geometric Mean (%GCV) were not calculated due to all Selumetinib plasma concentrations were below the level of detection at Cycle 2 Day 1. | NA (NA) — NA=Geometric Mean (%GCV) were not calculated due to all Selumetinib plasma concentrations were below the level of detection at Cycle 2 Day 1. | 2.05 (313.1)
  Selumetinib- Cycle 2 Day 14: number analyzed (Participants) | 2 | 1 | 7 | 12
  Selumetinib- Cycle 2 Day 14 | 72.5 (54.4) | 218 (NA) — Method of dispersion could not be reported for N<2 | 225 (82.6) | 283 (123.2)
  Selumetinib- Cycle 5 Day 1 | NA (NA) — NA=Geometric Mean (%GCV) were not calculated due to all Selumetinib plasma concentrations were below the level of detection at Cycle 5 Day 1. | NA (NA) — NA=Geometric Mean (%GCV) were not calculated due to all Selumetinib plasma concentrations were below the level of detection at Cycle 5 Day 1. | NA (NA) — NA=Geometric Mean (%GCV) were not calculated due to all Selumetinib plasma concentrations were below the level of detection at Cycle 5 Day 1. | NA (NA) — NA=Geometric Mean (%GCV) were not calculated due to all Selumetinib plasma concentrations were below the level of detection at Cycle 5 Day 1.
  Selumetinib- Cycle 5 Day 14: number analyzed (Participants) | 1 | 3 | 7 | 12
  Selumetinib- Cycle 5 Day 14 | 67.8 (NA) — Method of dispersion could not be reported for N<2 | NA (NA) — NA=Geometric Mean (%GCV) were not calculated due to all Selumetinib plasma concentrations were below the level of detection at Cycle 5 Day 14. | 529 (98.3) | 175 (192.7)

ADVERSE EVENTS:
Time Frame: From randomization through study completion data cutoff date of 28-June-2022 (Up to ~ 39 months)
Description: All-Cause Mortality (ACM): All allocated participants. Safety: All allocated participants who got ≥1 dose of study treatment. Per protocol, disease progression of cancer was not considered an AE unless related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" unrelated to study drug are excluded as AEs.
Arm/Group | Selumetinib 50mg + Pembrolizumab | Selumetinib 75mg + Pembrolizumab | Selumetinib 100mg + Pembrolizumab | Selumetinib 125mg + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 4/4 | 2/3 | 10/11 | 11/14
Serious Adverse Events (participants affected / at risk) | 2/4 | 2/3 | 4/11 | 4/14
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 11/11 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selumetinib 50mg + Pembrolizumab (N=4) | Selumetinib 75mg + Pembrolizumab (N=3) | Selumetinib 100mg + Pembrolizumab (N=11) | Selumetinib 125mg + Pembrolizumab (N=14)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selumetinib 50mg + Pembrolizumab (N=4) | Selumetinib 75mg + Pembrolizumab (N=3) | Selumetinib 100mg + Pembrolizumab (N=11) | Selumetinib 125mg + Pembrolizumab (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blindness (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Detachment of retinal pigment epithelium (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Visual field defect (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (4) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (4) | 4 (7) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fistula of small intestine (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (6) | 9 (9)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (6) | 7 (8)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2) | 7 (7) | 7 (7)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (5)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (1) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 7 (7) | 7 (8)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT03833427/Prot_SAP_000.pdf